CLINICAL TRIAL: NCT06418841
Title: A Prospective Observational Study Comparing Computer-Assisted Paramedian Approach Versus Conventional Midline Approach for Lumbar Puncture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChiCTR2300067936
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-02

CONDITIONS: Spinal Puncture
Keywords: computer modified paramedian approach technique, lumbar puncture, midline approach technique, puncture attempts, pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-Assisted Paramedian Approac Technique (Experimental): The L3-4 inter-laminar space will be selected as the target for puncture, and in the longitudinal direction, 1.0-1.5cm will be opened beside the upper edge of the spinous process (tip) of the lower vertebra as the entry point. The lumbar puncture needle will be inserted vertically along the axis of the anesthesia needle. The puncture path will be maintained completely perpendicular to the skin until the needle reached the PLTLF (posterior layer of the thoracolumbar fascia), where some resistance will be felt. The puncture direction is adjusted as needed. The tip of the needle will be tilted 20±10° in the sagittal direction and 15±5° inward such that the tip will point at the midpoint of the spinal canal. After the needle reaches the PLTLF, it will be further inserted 3-7 cm.
  Interventions: Procedure: Computer-Assisted Paramedian Approach Technique
- Conventional Midline Approach Technique (Experimental): Puncture will be performed on the posterior median line near the midpoint of the L3-4 Space of spinous process. The lumbar puncture needle will be inserted vertically along the axis of the anesthesia needle, or the tip of the needle will be tilted 15° in the sagittal direction toward the head, so that the needle path is parallel to the space of spinous process.
  Interventions: Procedure: Conventional Midline Approach Technique

INTERVENTIONS:
Procedure: Computer-Assisted Paramedian Approach Technique — Computer-Assisted Paramedian Approach Technique
  Arms: Computer-Assisted Paramedian Approac Technique
Procedure: Conventional Midline Approach Technique — Conventional Midline Approach Technique
  Arms: Conventional Midline Approach Technique

SUMMARY:
The goal of this clinical trial is to compare the effects of CMPAT and MAT in patients undergoing LP. Participants will be randomly assigned to either the CMPAT treatment group (group A) or the MAT treatment group (group B). Researchers will compare CMPAT treatment group and the MAT treatment group to see if the number of needle insertion attempts required for a successful LP, the puncture success rate, pain assessment in the back, head, and legs, and the occurrence of complications have different.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-99 years. Indication for lumber puncture (diagnostic lumbar puncture, analysis of cerebrospinal fluid composition, measurement of cerebrospinal fluid pressure, release of cerebrospinal fluid, lumbar cistern drain-age or intrathecal injection).

Body mass index between 18.5 and 35 kg/m2.

Exclusion Criteria:

* Cerebral hernia or known high cerebrospinal fluid pressure prone to cerebral hernia.
* Oral anticoagulant or antiplatelet therapy (≤3 days) or coagulation dysfunction, various factors lead to a higher risk of bleeding.
* Active infection or prior infection at the surgical site.
* Skin breakdown.
* Previous spine fusion surgery.
* Cauda equina syndrome.
* Pregnancy or breast feeding.
* Severe comorbid medical or psychiatric disorder.
* Unwilling to adhere to any of the required procedures.
* Cognitive impairment interfering with participant's ability to give full and - - informed consent or complete the baseline or follow-up assessments.
* Survival expectation less than 1 month.
* Moving abroad in 1 month.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of needle insertion attempts for successful LP | 30 minutes following treatment
  A successful puncture was defined as the presence of CSF outflow from the puncture needle. The number of needle insertion attempts was determined by the number of times the puncture needle was inserted into the target area.

SECONDARY OUTCOMES:
LP success rate | 30 minutes following treatment
  The parameters will measure the success rate of puncture in one attempt, the success rate of puncture within three attempts and the success rate of puncture within six attempts.
Assessment of back, head and leg pain using the NRS | before treatment, during surgery and 30 minutes,6 hours,1 days,3 days,7 days,2 weeks,4 weeks following treatment
  In the NRS, patients will be asked to indicate a number ranging from 0 to 10, which best reflects the intensity of their pain. A score of 0 indicates the absence of pain, while a score of 10 signifies the most excruciating pain imaginable. The NRS will be used to assess the severity of localised back pain, headaches, leg pain and numbness experienced by patients after LP.
Adverse events and other unintended effects | during surgery and 30 minutes,6 hours,1 days,3 days,7 days,2 weeks,4 weeks following treatment
  This study will monitor all adverse events during and after trial interventions, followed by causality assessment. In addition to risk mitigation protocols, we will remain vigilant about rare potential complications including drug allergies during anaesthesia; adjacent organ/ tissue injury; nerve, vascular or organ damage; paralysis, shock; difficulties/failures in puncture; needle breakage; persistent pain; neurological impairment; infections; CSF leakage; wound healing issues; epidural haematoma, etc. Their likelihood is extremely low under specialised surgical expertise.Any undesirable medical condition will be documented and reported transparently per ethics guidelines. The data safety monitoring board may recommend modifying/stopping the trial if safety concerns emerge. We will ensure diligent surveillance and injury precautions to safeguard participants.

OTHER OUTCOMES:
Locating time | 30 minutes following treatment
  The time taken to locate and mark the patient, defined as the duration from the beginning of positioning till the insertion of the anaesthetic needle.
Puncture time | 30 minutes following treatment
  The time taken to perform the LP defined as the duration from the first insertion of the puncture needle till the beginning of the outflow of CSF from the puncture needle.
Evaluation from physician | 30 minutes following treatment
  The methods for assessing LP immediately after physician evaluation are categorised as follows: very good, good, average, bad and very bad.
Evaluation from patient | 30 minutes following treatment
  Patient satisfaction, rated by patients immediately after LP, is classified as very good, good, average, bad or very bad.

IPD SHARING:
Plan to Share IPD: No